CLINICAL TRIAL: NCT04041271
Title: Jaw Kinematics and Muscle Activation in Patients With Non-specific Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: (717)108A-33
Record Dates: First submitted 2019-07-28; First posted 2019-08-01 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-09

CONDITIONS: Temporomandibular Disorder; Nonspecific Chronic Neck Pain; Biomechanical Phenomena
Keywords: Temporomandibular disorder; Nonspecific chronic neck pain; Jaw kinematics; Muscle activity; Muscle sensitivity; Forward head
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nonspecific chronic neck pain (NCNP) group: Subjects with nonspecific chronic neck pain will be included to perform clinical test and assess their jaw kinematics and muscle activation.
  Interventions: Other: Cervical range of motion (CROM); Other: Pressure pain threshold (PPT); Other: Cranial-cervical angle (CCA); Other: Jaw kinematics; Other: Muscle activation
- Control group: Healthy control subjects will be included to compare the differences in jaw kinematics, muscle activation and clinical tests between healthy subjects and subjects with nonspecific chronic neck pain. Subjects in this group will received the same assessment as the NCNP group.
  Interventions: Other: Cervical range of motion (CROM); Other: Pressure pain threshold (PPT); Other: Cranial-cervical angle (CCA); Other: Jaw kinematics; Other: Muscle activation

INTERVENTIONS:
Other: Cervical range of motion (CROM) — Subjects will perform full-range cervical flexion, extension, side-bending and rotation actively in sitting position. In supine position, cervical flexion-rotation will be performed passively by the assessor.
Other: Pressure pain threshold (PPT) — A digital algometer with rubber head will be used to apply pressure on the muscles of subjects. When the subjects start to feel pain, the algometer will be removed immediately.
Other: Cranial-cervical angle (CCA) — Subjects will stand in a relaxed position with colour markers on the earlobe and C7 spinous process. A photo of the head posture will be taken to calculate the included angle between the markers and the horizontal line.
Other: Jaw kinematics — Jaw kinematics is measured by Ultrasonic Jaw Motion Analyzer (Zebris). The subjects will perform jaw opening, closing, lateral left, lateral right and protrusion for three times.
Other: Muscle activation — Surface electromyography is used to assess the activities of bilateral masseter, anterior temporalis, sternocleidomastoid muscle and upper trapezius. Subjects will perform jaw resting and clenching.

SUMMARY:
Temporomandibular disorder (TMD) is a collective term for pain and dysfunction of the masticatory muscles and temporomandibular joint (TMJ). Typical signs and symptoms of TMD includes regional pain, noises from the TMJs and limitations in jaw movements. Altered jaw kinematics and muscle activity have also been reported. TMD may be related to neck problems. Over 50% of patients with TMD suffer from nonspecific neck pain. Patients with TMD often have symptoms over neck, including upper cervical spine movement impairment and reduced cervical muscles endurance. Conversely, TMD may also develop in patients with neck pain. Twenty to thirty-three percent of patients with neck pain also have TMD. Subjects with neck pain present with a twofold higher prevalence of TMD than those without neck pain. In patients with neck pain, the development or perpetuation of TMD may be due to the anatomical connection between TMJ and neck: neck posture affects the mandible position and sensory inputs from the cervical-mandibular region converge at the trigemino-cervical nucleus. Early identification of TMD is essential but to our knowledge, no study has investigated whether patients with neck pain demonstrate altered jaw movement and muscle activity, which is associated with TMD. The purposes of this proposal are to compare the jaw kinematics, muscle activity and muscle sensitivity in healthy individuals and patients with non-specific chronic neck pain (NCNP). This study also aimed to investigate the relationship between forward-head posture and the jaw kinematics, muscle activity as well as muscle sensitivity. With a cross-sectional exploratory study design, 30 healthy control subjects and 30 subjects with NCNP will be recruited. Clinical assessments will include cervical range of motion (CROM), pressure pain threshold (PPT) over the cervical-mandibular region and the cranial-cervical angle (CCA). Jaw kinematics will be measured by Ultrasonic Jaw Motion Analyzer (Zebris GmbH) during functional jaw movements. Muscle activities are record from bilateral anterior temporalis, masseter, sternocleidomastoid muscle and upper trapezius by surface electromyography during resting and clenching.

ELIGIBILITY:
Inclusion Criteria (nonspecific chronic neck pain group):

* Aged between 20 to 65 years old
* Mechanical pain that provoked by sustained neck postures or specific neck movements without any identifiable diseases or structure anomalies
* Chronic or recurrent neck pain of at least 3 months duration
* Minimum of 3 points on the numerical pain rating scale (NPRS) over cervical region
* Without any pain, clicking or range of motion limitation over TMJ

Inclusion Criteria (healthy control group):

* Age (± 5 years) and gender match to NCNP group
* No pain or clinical pathology involving the masticatory system or cervical spine for at least one year prior to the start of the study

Exclusion Criteria (both groups):

* Serious injury, tumor, infection
* Recent cervical-cranial surgery
* Neurologic involvement
* Inflammatory rheumatic diseases
* Pregnancy
* Nonmechanical cause of neck pain (e.g. herniated disk, spinal fractures)
* Had been diagnosed with spinal conditions (e.g. spondylolisthesis)
* Shoulder pain within 1 years
* Loss of posterior tooth
* Dental pain or periodontal problems
* Orthodontic, orofacial myofunctional or TMD treatment within 3 months
* Use of analgesic or anti-inﬂammatory drugs within 3 days

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with nonspecific chronic neck pain for at least 3 months and the matched healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Jaw maximum range of motion | Immediately during the experiment
  Including maximum mouth opening, lateral right, lateral left, and protrusion, which will be described with millimeter (mm)
Jaw velocity | Immediately during the experiment
  Jaw opening and closing velocity, which will be described with millimeter per second (mm/s)
Condylar rotation | Immediately during the experiment
  The rotation will be described with degree (°).
Condylar translation | Immediately during the experiment
  Including condylar translation and condylar path length, which will be described with millimeter (mm)
Muscle activation | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the masseter, anterior temporalis, sternocleidomastoid muscle and upper trapezius will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %).

SECONDARY OUTCOMES:
Cervical and jaw range of motion | Immediately during the experiment
  Including range of motion of cervical flexion, cervical extension, cervical side-bending,cervical rotation and cervical flexion-rotation as well as maximum mouth opening, jaw lateral right, jaw lateral left, protrusion. The motion will be described with degree (°).
Pressure pain threshold | Immediately during the experiment
  Pressure pain threshold of masseter, anterior temporalis, sternocleidomastoid muscle, upper trapezius and suboccipitals will each be averaged and will be described with kg/cm2.
Cranial-cervical angle | Immediately during the experiment
  Cranial-cervical angle will be measured as the included angle between the ear lobe, C7 spinous process and the horizontal line and will be described with degree (°).

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan